CLINICAL TRIAL: NCT00644436
Title: A Study of the Substantivity of Tetrix Cream
Brief Title: Study to Determine if Tetrix Cream is Removed From the Hands by Gentle Washing With Soap and Water
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Coria Laboratories, Ltd. (Industry)
Responsible Party: David Innes Cargill, PhD, Coria Laboratories
Allocation: Randomized | Model: Single Group | Masking: Single
Other Study IDs: 806 805 09 001
Record Dates: First submitted 2008-03-20; First posted 2008-03-26 (Estimated); Last update posted 2008-03-28 (Estimated); Status verified 2008-03

CONDITIONS: Healthy
Keywords: tetrix cream; substantivity; resistance to a gentle wash; Tetrix Cream remaining on hands after gentle washing with soap and water.

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Single topical application
  Interventions: Device: Tetrix
- 2 (Active Comparator): Single topical application
  Interventions: Device: Tetrix

INTERVENTIONS:
Device: Tetrix — single topical application
  Arms: 1
Device: Tetrix — Single topical application
  Arms: 2

SUMMARY:
To determine if Tetrix Cream remains on the hands after gentle washing with soap and water

ELIGIBILITY:
Inclusion Criteria:

* Normal subjects
* Male and Female

Exclusion Criteria:

* Under the age of 18 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2007-11; Primary Completion 2007-11 (Actual); Study Completion 2007-11 (Actual)

PRIMARY OUTCOMES:
amount of Tetrix remaining on the skin compared to control, after gentle washing with soap | 30 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Zoe Draelos, MD, Principal Investigator — Dermatology Consulting Service
Locations (1):
- Dermatology Consulting Services, High Point, South Carolina, United States